CLINICAL TRIAL: NCT02128477
Title: Predictive Value of Periodic Repolarization Dynamics in Post-Infarction Patients: Validation Study
Brief Title: Predictive Value of Periodic Repolarization Dynamics in Post-Infarction Patients
Acronym: PRD-MI
Status: Completed | Type: Observational
Sponsor: Thebiosignals.com (Other)
Responsible Party: Sponsor
Other Study IDs: BIO012014
Record Dates: First submitted 2014-02-05; First posted 2014-05-01 (Estimated); Last update posted 2017-01-25 (Estimated); Status verified 2017-01

CONDITIONS: Myocardial Infarction
Keywords: Myocardial infarction; Repolarization instability; Ventricular fibrillation
MeSH Terms: conditions — Myocardial Infarction; Ventricular Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Increased periodic repolarization dynamics (PRD) indicate increased risk of death in cardiac patients. This study thoughts to prospectively validate the prognostic value of PRD in post-infarction patients.

DETAILED DESCRIPTION:
Periodic repolarization dynamics (PRD) reflect periodic changes of repolarization instability located in the low-frequency spectral range. Level of PRD can be assessed using a high resolution surface ECG recorded in the 12-leads of Frank leads configuration during resting conditions.

Increased levels of PRD have been associated with sympathetic overactivity and increased risk of mortality in survivors of acute myocardial infarction and patients undergoing a clinically indicated exercise test.

ELIGIBILITY:
Inclusion Criteria:

* previous myocardial infarction >4 weeks
* age >18 years

Exclusion Criteria:

* life expectancy < 1 year due to non-cardiac causes
* unable to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: myocardial infarction
Sampling Method: Probability Sample
Enrollment: 754 (Actual)
Dates: Start 2010-10 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Number of total deaths | 24 months

SECONDARY OUTCOMES:
Number of cardiovascular deaths | 24 months

CONTACTS AND LOCATIONS:
Locations (1):
- Eberhard-Karls-University Tuebingen, Tübingen, Baden-Wurttemberg, Germany